CLINICAL TRIAL: NCT06166342
Title: Efficacy Evaluation of TCI153 Probiotics for Skin Beautification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23-091-B
Record Dates: First submitted 2023-11-29; First posted 2023-12-12 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo sachet (Placebo Comparator): consume 1 sachet per day
  Interventions: Dietary Supplement: Placebo sachet
- TCI153 sachet (Experimental): consume 1 sachet per day
  Interventions: Dietary Supplement: TCI153 probiotic sachet

INTERVENTIONS:
Dietary Supplement: Placebo sachet — Consume 1 sachet daily
  Arms: Placebo sachet
Dietary Supplement: TCI153 probiotic sachet — Consume 1 sachet daily
  Other Names: Ligilactobacillus salivarius TCI153 sachet
  Arms: TCI153 sachet

SUMMARY:
To assess TCI153 prebiotics product on skin condition improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 18 years old

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* Patients with diseases of the skin, liver, kidney.
* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Received facial laser therapy, chemical peeling or UV overexposure (> 3 hr/week) in the past 4 weeks.
* Constant drug use
* Students who are currently taking courses taught by the principal investigator of this trial.
* Subject who is not willing to have their photos published in public.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
The change of skin wrinkles | Change from Baseline skin wrinkles at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin wrinkles. Units: arbitrary units
The change of skin texture | Change from Baseline skin texture at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin melanin index | Change from Baseline skin melanin index at 8 weeks
  Mexameter® MX18 was utilized to measure skin melanin index. Units: arbitrary units
The change of skin L* value | Change from Baseline L* value at 8 weeks
  Chroma Meter MM500 was utilized to measure skin L* value. Units: arbitrary units, 0-100

SECONDARY OUTCOMES:
The change of skin elasticity | Change from Baseline skin elasticity at 8 weeks
  Cutometer® MPA580 was utilized to measure skin elasticity. Units: arbitrary units
The change of skin erythema index | Change from Baseline skin erythema index at 8 weeks
  Mexameter® MX18 was utilized to measure skin erythema index. Units: arbitrary units
The change of skin moisture | Change from Baseline skin moisture at 8 weeks
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
The change of transepidermal water loss (TEWL) | Change from Baseline TEWL at 8 weeks
  Tewameter® TM 210 was utilized to measure TEWL. Units: g/hm²
The change of skin pores | Change from Baseline AGEs at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin pores. Units: arbitrary units
The change of gut microbiome composition | Change from Baseline AGEs at 8 weeks
  Gut microbiome sequencing

OTHER OUTCOMES:
The change of liver function biomarkers (AST, ALT) of blood | Change from Baseline liver function biomarkers at 8 weeks
  Fasting venous blood was sampled to measure liver function biomarkers
The change of renal function biomarkers (creatinine, BUN) of blood | Change from Baseline renal function biomarkers at 8 weeks
  Fasting venous blood was sampled to measure renal function biomarkers
The change of fasting blood glucose | Change from Baseline blood glucose at 8 weeks
  Fasting venous blood was sampled to measure blood glucose
The change of sialic acid | Change from Baseline sialic acid at 8 weeks
  Fasting venous blood was sampled to measure sialic acid
The change of Epidermal Growth Factor (EGF) | Change from Baseline EGF at 8 weeks
  Fasting venous blood was sampled to measure EGF

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy & Science, Tainan, Taiwan